CLINICAL TRIAL: NCT01038271
Title: A Randomized, Controlled Trial of Integrated vs. Standard Palliative Care in Patients With Advanced NSCLC
Brief Title: Integrated Versus Standard Palliative Care in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Thoracic Oncology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-030
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: palliative care
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Palliative Care Group (Active Comparator)
  Interventions: Other: Standard Palliative Care Group
- Integrated Palliative Care Group (Active Comparator)
  Interventions: Other: Integrated Palliative Care Intervention

INTERVENTIONS:
Other: Standard Palliative Care Group — Participant is referred to the Palliative Care Team at any time.
  Arms: Standard Palliative Care Group
Other: Integrated Palliative Care Intervention — Participant meets with the Palliative Care Team within 3 weeks of being randomized
  Arms: Integrated Palliative Care Group

SUMMARY:
The main purpose of this study is to compare two types of treatment-standard palliative care (which usually is given towards the end of life) and integrated palliative care (which is given soon after diagnosis) to see which is better for improving quality of life of participants with advanced non-small cell lung cancer. Palliative care is care that tries to lessen the symptoms of a disease. Although many people with advanced lung cancer receive palliative care or hospice toward the end of their disease, the entire course of their disease is often complicated by physical and emotional difficulties. Palliative care may be useful when it is started soon after diagnosis.

DETAILED DESCRIPTION:
* Participants with advanced small-cell lung cancer, will be asked to fill out some quality of life questionnaires that help to measure their quality of life (QOL), mood and understanding of their illness. They will also be asked to identify an important person in their life, either a relative or friend, who they count on for help and support. The research staff will contact that individual and ask them to if they want to participate in the caregiver part of this study.
* Lung cancer participants will then be randomized into one of the two study groups: integrated palliative care or standard palliative care.
* Participants assigned to the Standard palliative care group will be referred to the Palliative Care Team at their doctor's or their request at any time. At that time the Palliative Care Team (PCT) will follow and treat the participant as they would any other cancer patient. Research staff will request the participant to fill out QOL, mood & illness understanding questionnaires about 12, 18 and 24 weeks after they sign the consent form. Their caregiver will be asked to fill out the FamCare form at 12, 18 and 24 weeks.
* Participants assigned to the Integrated Palliative Care group will have an appointment with the Palliative Care Team within 3 weeks of being randomized. The palliative care physician will formulate a care plan based on the participant's and caregiver's issues and needs. The PCT will meet with the participant on a regular basis, a minimum of every 6 weeks. These visits wil vary with the participant's needs and may include individual or group meetings with the physicians, nurse practitioners, social workers or chaplains. Research staff will ask you to fill out QOL, mood & illness understanding questionnaires about 12, 18 and 24 weeks after they sign the consent form. Their caregiver will be asked to fill out the FamCare form at 12, 18 and 24 weeks.
* Participants will be in this research study for about 24 weeks or 6 months. After this 6 month period is over, care by the Palliative Care Team my continue but the participants will not be asked to fill out more questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed incurable NSCLC, stage IIIB with a pleural or pericardial effusion or stage IV
* Performance status 0-2
* Diagnosis of advanced NSCLC within the previous eight weeks
* Ability to read and respond to questions in English
* Permission of attending physician

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* Existence of other co-morbid disease, which in the opinion of the investigator prohibits participation in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Assess the impact of early integration with palliative care on QOL in patients with advanced NSCLC. | 3 years

SECONDARY OUTCOMES:
Assess the impact of early integration with palliative care on mood and illness understanding. | 3 years
Assess the impact of early integration with palliative care on family caregiver satisfaction, mood, and QOL both during care and after death. | 3 years
Compare hospice referrals and length of stay on hospice between study arms. | 3 years
Compare outpatient code status documentation between study arms. | 3 years
Compare the percentage of patients on each arm who received chemotherapy within one month of death. | 3 years
Determine the amount of time palliative care devotes to illness understanding, symptom management, decision-making, and coping with an illness in the outpatient setting. | 3 years
Health Care Costs | After death
  We will utilize the hospital cost accounting/billing system to determine health care costs as per study arm

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Result] Jacobsen J, Jackson V, Dahlin C, Greer J, Perez-Cruz P, Billings JA, Pirl W, Temel J. Components of early outpatient palliative care consultation in patients with metastatic nonsmall cell lung cancer. J Palliat Med. 2011 Apr;14(4):459-64. doi: 10.1089/jpm.2010.0382. Epub 2011 Mar 18. PMID 21417739
- [Result] Temel JS, Greer JA, Admane S, Gallagher ER, Jackson VA, Lynch TJ, Lennes IT, Dahlin CM, Pirl WF. Longitudinal perceptions of prognosis and goals of therapy in patients with metastatic non-small-cell lung cancer: results of a randomized study of early palliative care. J Clin Oncol. 2011 Jun 10;29(17):2319-26. doi: 10.1200/JCO.2010.32.4459. Epub 2011 May 9. PMID 21555700
- [Result] Greer JA, Pirl WF, Jackson VA, Muzikansky A, Lennes IT, Heist RS, Gallagher ER, Temel JS. Effect of early palliative care on chemotherapy use and end-of-life care in patients with metastatic non-small-cell lung cancer. J Clin Oncol. 2012 Feb 1;30(4):394-400. doi: 10.1200/JCO.2011.35.7996. Epub 2011 Dec 27. PMID 22203758
- [Result] Pirl WF, Greer JA, Traeger L, Jackson V, Lennes IT, Gallagher ER, Perez-Cruz P, Heist RS, Temel JS. Depression and survival in metastatic non-small-cell lung cancer: effects of early palliative care. J Clin Oncol. 2012 Apr 20;30(12):1310-5. doi: 10.1200/JCO.2011.38.3166. Epub 2012 Mar 19. PMID 22430269
- [Result] Yoong J, Park ER, Greer JA, Jackson VA, Gallagher ER, Pirl WF, Back AL, Temel JS. Early palliative care in advanced lung cancer: a qualitative study. JAMA Intern Med. 2013 Feb 25;173(4):283-90. doi: 10.1001/jamainternmed.2013.1874. PMID 23358690